CLINICAL TRIAL: NCT02162381
Title: Methylphenidate Effect on Performing Humphrey Visual Fields
Brief Title: Methylphenidate Effect on Humphrey Visual Fields
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Bialer, Dr. Omer Y. Bialer, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0105-14-RMC
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Visual Field Tests
Keywords: Humphrey visual fields; methylphenidate; attention deficit disorder; MoCa questionnaire
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylphenidate provided (Experimental): the study group will be given a single pill containing methylphenidate 10mg to be taken 2 hours before their visual field test
  Interventions: Drug: methylphenidate; Other: guidance
- control (Active Comparator): control group will not be given any placebo and will perform a repeat visual field testing without any prior preparation
  Interventions: Other: guidance

INTERVENTIONS:
Drug: methylphenidate — a single dose of methylphenidate 10 mg to be taken orally in the morning
  Other Names: Ritalin
  Arms: methylphenidate provided
Other: guidance — subjects will be given an explanation and advice about how to perform well in visual field testing

SUMMARY:
Study will include adults with abnormal visual fields. Half of them will be given either methylphenidate 10mg 2 hours before repeating the visual field test. the rest will serve as controls. All Subjects will also have a complete eye examination, a short questionnaire and a questionnaire to screen for attention deficit disorder. The investigators will compare the visual field results between the 2 tests.

DETAILED DESCRIPTION:
Healthy adults with abnormal visual fields will be offered to participate Subjects will have a complete ophthalmic examination including dilated fundus examination.

Subjects with clear explanation for a visual field defect (e.g. optic neuropathy or retinal disorder) will be excluded from the study the subjects will be randomly assigned to the study group and control group using a 1:1 allocation.

Subjects in the study group will be provided with a single tablet of methylphenidate 10 mg to be taken orally 2 hours before repeating their visual field test.

The control group will not receive any placebo Both groups will repeat their visual fields. Both groups will fill out a short questionnaire to evaluate their experience in the second visual field test.

The study group will also fill out a screening questionnaire to rule out previously undiagnosed attention deficit disorder.

Two experienced ophthalmologists will separately interpret the visual fields results and compare the first and second visual fields of each subject, while being blinded to which group he was in.

Subjects will be provided with their test results and the ophthalmologist interpretation.

ELIGIBILITY:
Inclusion Criteria:

* abnormal visual fields
* must be able to swallow pills

Exclusion Criteria:

* psychiatric disorder
* dementia
* ocular disorder which is known to cause abnormal visual fields
* prescription of psychoactive medications
* visual acuity lower than 20/100
* cardiac arrhythmia
* hypersensitivity to methylphenidate
* prescription of warfarin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06; Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
improvement rate of a repeat visual field result | immediate
  the percentage of subjects whose second (repeat) visual field has improved compared to the first visual field - as interpreted by independent blinded ophthalmologists

SECONDARY OUTCOMES:
Humphrey visual field Mean Deviation (MD) | immediate
  the MD of the Humphrey visual field in the study and control groups will be compared
Humphrey visual field severity score | immediate
  based on the Humphrey visual field gray scale each visual field will be given a score between 1 and 4. 1 = normal 2=enlargement of the blind spot 3=either a nasal or temporal visual field 4= diffuse visual field loss

CONTACTS AND LOCATIONS:
Overall Officials: Omer Y Bialer, M.D., Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center - Beilinson campus, Petah Tikva, Israel

REFERENCES:
- [Background] Martin L, Aring E, Landgren M, Hellstrom A, Andersson Gronlund M. Visual fields in children with attention-deficit / hyperactivity disorder before and after treatment with stimulants. Acta Ophthalmol. 2008 May;86(3):259-64. doi: 10.1111/j.1755-3768.2008.01189.x. PMID 18494726
- [Background] Challman TD, Lipsky JJ. Methylphenidate: its pharmacology and uses. Mayo Clin Proc. 2000 Jul;75(7):711-21. doi: 10.4065/75.7.711. PMID 10907387
- [Background] Dodson WW. Pharmacotherapy of adult ADHD. J Clin Psychol. 2005 May;61(5):589-606. doi: 10.1002/jclp.20122. PMID 15723384
- [Derived] Sternfeld A, Bialer OY, Keidar D, Megiddo E, Budnik I, Stiebel-Kalish H, Livnat T. A Single Low-Dose of Methylphenidate Improves Abnormal Visual Field Testing. Curr Eye Res. 2021 Aug;46(8):1232-1239. doi: 10.1080/02713683.2020.1858430. Epub 2020 Dec 21. PMID 33342320